CLINICAL TRIAL: NCT03566888
Title: Validation of a Noninvasive Automated Blood Pressure Device
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Todd Schroeder, Assistant Professor, University of Southern California
Other Study IDs: HS-17-00139
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single Group: 85 eligible study participants
  Interventions: Device: Blood pressure assessment

INTERVENTIONS:
Device: Blood pressure assessment — Validation of an automated blood pressure device

SUMMARY:
The investigator's objective is to validate the novel automated blood pressure device against the requirements set forth in the AAMI_ISO 81060-2:2010 standard in voluntarily consented study participants.

DETAILED DESCRIPTION:
A new prototype blood pressure cuff has been designed for the higi SH llc health stations. This new cuff accurately captures blood pressure (BP) by emulating a fitted cuff which is used in conjunction with a mercury sphygmomanometer, the accepted gold standard for measuring BP values in most clinical facilities. The cuff is driven by a motor and gearhead to automatically "wrap" the cuff around a user's arm when they initiate a BP test. A BP measurement is then taken by an Original Equipment Manufacturer (OEM) BP module using an algorithm developed for use with a fitted cuff; the same module one would expect to find in a clinic or doctor's office. For the device to pass the AAMI_ISO 81060-2:2010 standard statistical requirements and thus, be considered a valid device for measuring BP it will need to meet the standards criteria 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 12 to 92 years of age.
* generally healthy but can be on medication for blood pressure regulation.

Exclusion Criteria:

* heart disease is present such as, coronary artery disease, cardiomegaly, irregular heart rhythm, atrial fibrillation, heart valve disease, congenital heart disease, cardiomyopathy, pericardial effusion, Marfan syndrome, and heart murmurs.
* using a pacemaker to maintain a suitable heart rate.
* missing their natural left arm.
* exhibit a musculoskeletal disorder that may prevent them from sitting upright for a period of time (~40min) or prevent a BP reading taken from the left arm.
* Special populations, for example pregnant women and patients with known arrhythmias.

Ages: 12 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals between the ages of 12-92 years, generally healthy, and have not been diagnosed with heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Systolic and Diastolic blood pressure (criteria 1 and 2) | 60 minutes
  Mean value of the differences of the paired (i.e., device under test - reference method) determinations for all study participants shall be within or equal to ± 5 mmHg with a standard deviation no greater than 8 mmHg (criterion 1). Standard deviation of the averaged paired determinations per participant shall meet the criterion 2 listed in the standard.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schroeder, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No